CLINICAL TRIAL: NCT04188197
Title: Assisting Smokers to Switch to a JUUL E-Cigarette by Devaluing Combustible Cigarettes
Acronym: RECON
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rose Research Center, LLC (Industry)
Collaborators: Foundation for a Smoke Free World INC (Other)
Responsible Party: Principal Investigator, Jed Rose, President and CEO, Rose Research Center, LLC
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RECON
Record Dates: First submitted 2019-09-09; First posted 2019-12-05 (Actual); Results first posted 2025-04-20 (Actual); Last update posted 2025-04-20 (Actual); Status verified 2025-04

CONDITIONS: Smoking Cessation; Harm Reduction; E-Cig Use; Cigarette Smoking; Tobacco Dependence; Tobacco Use Cessation
MeSH Terms: conditions — Smoking Cessation; Harm Reduction; Vaping; Cigarette Smoking; Tobacco Use Disorder; Tobacco Use Cessation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- e-Cigarette Matched to Usual Brand Cigarette (Experimental): JUUL and cigarette flavor matched ("Mint" for menthol smokers and "Virginia Tobacco" for non-menthol smokers);
  Interventions: Other: JUUL
- e-Cigarette Unmatched to Usual Brand Cigarette (Experimental): JUUL and cigarette flavor unmatched ("Virginia Tobacco" for menthol smokers and "Mint" for non-menthol smokers).
  Interventions: Other: JUUL

INTERVENTIONS:
Other: JUUL — Subjects will be instructed to use the JUUL as often as they like during the 12-week product use period. They will also be instructed to use JUUL immediately before each cigarette to relieve their craving as much as possible before smoking their usual brand. The JUUL will also be the first product that they are instructed to use each morning. Smokers will be told to try to completely substitute JUUL for cigarettes by the end of the first week of use.

SUMMARY:
This study will evaluate a reward devaluation strategy in which smokers use the JUUL e-cigarette immediately before any combustible cigarettes (CCs) are smoked. This procedure is predicted to accomplish three goals: 1) the rewarding effects of CC will be disrupted because subjects will already have attained fairly high peak nicotine concentrations immediately before smoking the cigarette. This reduces the rewarding effect of smoking, in part from receptor desensitization that occurs following nicotine exposure, which reduces the response to a subsequent dose of nicotine, and in part from satiating the drive to smoke; 2) the use of the JUUL will become associated with the same cues that elicit smoking, thereby promoting the substitution of JUUL use for CC use; and 3) ad libitum nicotine intake from the JUUL and its rewarding effects will be maximized because, unlike CC, they will be experienced after a period of nicotine deprivation. Thus, despite a lower per-puff nicotine dose relative to CC, the pharmacologic impact and reinforcing effect will be maximized. The study will evaluate two flavors (Mint and Virginia Tobacco), randomly assigned, to determine if flavor assignment (similar to the subjects' usual brand of CC or different than the subjects usual brand CC) has an effect on the success of this reconditioning procedure.

ELIGIBILITY:
Inclusion Criteria:

1. Has signed the ICF and is able to understand the information provided in the ICF.
2. Is 21 to 65 years of age (inclusive) at screening.
3. Smokes ≥ 10 commercially available CCs per day (no brand restrictions), for the last 12 months.
4. Expired air CO reading of at least 10 ppm as assessed at the screening session.
5. Interested in switching to an electronic cigarette.
6. Willing and able to comply with the requirements of the study.
7. Owns a smartphone with text message and data capabilities compatible with necessary surveys.

Exclusion Criteria:

1. Is unhealthy or cannot participate in the study for any reason (e.g., medical, psychiatric, and/or social reason) as judged by the Investigator or designated medical staff based on all available assessments from the screening period (e.g., safety laboratory, vital signs, physical examination, ECG, concomitant medications and medical history).
2. PHQ-9 score greater than 9, or a score greater than 0 on item #9 ("Thoughts that you would be better off dead, or of hurting yourself in some way") at screening.
3. Planned use of an FDA-approved smoking cessation product during the study.
4. High Blood Pressure (systolic >150 mm Hg, diastolic >95 mm Hg) at screening.
5. Body mass index (BMI) less than 15.0 kg/m2 or greater than 40.0 kg/m2.
6. Coronary heart disease, structural cardiac disease (including, but not limited to valvular heart disease or cardiac murmurs), cardiac dysrhythmias, syncope, cardiac chest pain, or history of heart attack or heart failure.
7. Has received psychotherapy or behavioral treatments within 30 days of screening, or during the study.
8. Taking antidepressants or psychoactive medications (e.g. antipsychotics, benzodiazepines, hypnotics).
9. Use of any of these products in the past 30 days:

   1. Illegal drugs (or if the urine drug screen is positive for cocaine, THC, amphetamines, methamphetamines, or opiates);
   2. Experimental (investigational) drugs that are unknown to the subject;
   3. Chronic opiate use.
10. Use of smokeless tobacco (chewing tobacco, snuff), cigars (except for "Black & Mild" cigars or Cigarillos), pipes, hookah, e-cigarettes, nicotine replacement therapy or other smoking cessation treatments within 14 days of screening.
11. Pregnant or nursing (by self-report) or positive pregnancy test.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2019-08-26 (Actual); Primary Completion 2021-03-02 (Actual); Study Completion 2021-06-22 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Rose Research Center, Charlotte, North Carolina
  - Rose Research Center, Raleigh, North Carolina

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First participant was consented on 26-Aug-2019, final participant was consented on 20-Nov-2020.
Period: Overall Study
Arm/Group | e-Cigarette Matched to Usual Brand Cigarette | e-Cigarette Unmatched to Usual Brand Cigarette
Started | 25 | 25
Completed | 20 | 22
Not Completed | 5 | 3
Not completed — Lost to Follow-up | 4 | 1
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Pregnancy | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | e-Cigarette Matched to Usual Brand Cigarette | e-Cigarette Unmatched to Usual Brand Cigarette | Total
Number analyzed (Participants) | 25 | 25 | 50
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 25 | 25 | 50
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 46 (9.51) | 46 (11.82) | 46 (10.72)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 14 | 23
  Male | 16 | 11 | 27
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 4 | 5
  Not Hispanic or Latino | 24 | 21 | 45
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 6 | 6 | 12
  White | 19 | 19 | 38
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 25 | 25 | 50

OUTCOME MEASURES:

1. Primary Outcome: Effects of Devaluation on Switching From Cigarettes to the JUUL E-cigarette
Description: Biochemically verified smoking abstinence during weeks 9-12, i.e., self-report of no smoking confirmed by an expired air CO reading of <5 ppm.
Time Frame: During Weeks 9-12
Measure: Count of Participants; unit: Participants
Arm/Group | e-Cigarette Matched to Usual Brand Cigarette | e-Cigarette Unmatched to Usual Brand Cigarette
Number analyzed (Participants) | 25 | 25
Participants | 4 | 4

2. Secondary Outcome: Changes in Cigarette Reward With Subsequent Switching Behavior
Description: Characterize changes in the two primary scales of the Cigarette Evaluation Questionnaire (mCEQ), assessing smoking satisfaction and psychological reward, over the first week of the study period. The mCEQ uses a 7-point scale (0=Not at all; 1=Very little; 2=A little; 3=Moderately; 4=A lot, 5=Quite a lot; 6=Extremely) to measure all subscales: Satisfaction, Psychological Reward, Enjoyment of Respiratory Tract Sensations, Craving Reduction, Aversion. Both subscales have the same "7-point scale" range.
Time Frame: Week 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | e-Cigarette Matched to Usual Brand Cigarette | e-Cigarette Unmatched to Usual Brand Cigarette
Number analyzed (Participants) | 25 | 25
score on a scale
  Change in Satisfaction scale of mCEQ at 1 week (V3) minus baseline (V2) | -0.8 (1.0) | -0.8 (1.2)
  Change in Psych Reward scale of mCEQ at 1 week (V3) minus baseline (V2) | -0.1 (1.1) | -0.4 (0.9)

ADVERSE EVENTS:
Time Frame: 12 weeks
Arm/Group | e-Cigarette Matched to Usual Brand Cigarette | e-Cigarette Unmatched to Usual Brand Cigarette
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/25
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/25
Other Adverse Events (participants affected / at risk) | 13/25 | 14/25
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | e-Cigarette Matched to Usual Brand Cigarette (N=25) | e-Cigarette Unmatched to Usual Brand Cigarette (N=25)
Cough (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 7 (8)
Upper Respiratory Infection (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 6 (6)
Headache (Nervous system disorders) | 1 (1) | 5 (5)
Nausea (Nervous system disorders) | 2 (2) | 1 (1)
Elevated Blood Pressure (Cardiac disorders) | 2 (2) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-09-29): https://cdn.clinicaltrials.gov/large-docs/97/NCT04188197/Prot_SAP_000.pdf